CLINICAL TRIAL: NCT01746433
Title: Evaluation of the Mobility of Elderly Patients (> 65 Years) When Using the "l'Ergonome" Mobility Device: a Randomized, Monocentric Study
Brief Title: Mobility of Elderly Patients When Using the "l'Ergonome" Mobility Device
Acronym: L'ERGONOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LOCAL/2012/EVFN-02; 2012-A01141-42 (Other: RCB number)
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Supine Position; Elderly
MeSH Terms: conditions — Deception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hanging Triangle Bar (Active Comparator): The patients randomized to this group will use a hanging triangle bar for aid in sitting up exercises.
  No particular brand of hanging bar is targeted.
  Interventions: Other: Sitting up
- Ergonome (Experimental): The patients randomized to this group will use the "l'ERGONOME" device for aid in sitting up exercises.
  Commercial name of the device: SAM ERGONOM (TM)
  Manufacturer: Medicatlantic groupe Winncare, Le Pas du Château, 85680 Saint-Paul-Mont-Penit
  Interventions: Other: Sitting up

INTERVENTIONS:
Other: Sitting up — The patient is positioned on a Winncare type bed dressed with a pressure-sensor sheet and equipped with either a hanging triangle bar (supporting arm of the bar is adjusted to 30 degrees) or an ERGONOME device according to randomization.
  The patient is first installed on the bed in a strictly supine position, the pelvis centered, and the greater trochanter over the fold of the backrest.
  The investigator then gives instructions on how to use the randomized device (correct hand placement).
  The patient is asked to sit up twice (two consecutive attempts). The first attempt is a learning attempt. The observations necessary for this study will be taken on the second attempt. Thus the second sitting attempt is timed, video-taped and recorded via the pressure-sensor sheet beneath the patient.

SUMMARY:
The main objective of this study is to compare the percentage of patients that successfully pass from a laying position to a sitting position in less than 10 seconds between study arms:

* experimental arm: these patients will use the ERGONOME device to help them sit up
* standard arm: these patients will use traditional hanging triangle bar to help them sit up

DETAILED DESCRIPTION:
The secondary objectives of this study are to compare the following between study arms:

* The average time (s) required to sit up
* How the patient's center of gravity moves in relation to a fixed axis

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient must be in stable medical condition (no complications for the last 10 days)
* The patient is incapable of changing from a laying position to a sitting position by his/herself in <10 secondes, and requires help for such movement
* The patient has a sitting-balance score > 2/4 (Brun et al 1991: Actual Rééduc Réadaptat: (16):412-7))

Exclusion Criteria:

* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient has fractured vertebrae or pelvis
* The patient has a weak heart
* The patient has joint pain localized to the dorso-lumbar region
* The patient has behavioral disorders (opposition, agitation, dementia)
* The patient has a medical prescription for physical restraint by bed rails.
* The patient is incapable of understanding the utility of the proposed technical aide, and using it for rolling and sitting up (notion of compliance).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Successful transition from a laying position to a sitting position | Baseline (day 0)
  yes/no

SECONDARY OUTCOMES:
Time needed to sit up | baseline (day 0)
  (minutes)
  The time needed to sit up is defined as follows:
  * The minimum time recorded for two attempts in the "Hanging Triangle Bar" group
  * The maximum time recorded for two attempts in the "Ergonome group"
Shift in the patient's center of mass (cm) | baseline (day 0)
  Shift in the patient's center of mass away from the x-axis of a pressure-sheet placed on the bed.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Viollet, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France